CLINICAL TRIAL: NCT01106313
Title: Insulin Resistance in Patients With Major Depression
Status: Completed | Type: Observational
Sponsor: Stanford University (Other)
Collaborators: American Diabetes Association (Other)
Responsible Party: Principal Investigator, Natalie Rasgon, Principal Investigator, Stanford University
Other Study IDs: SU-02172010-5003; eProtocol 17089
Record Dates: First submitted 2010-04-16; First posted 2010-04-19 (Estimated); Last update posted 2017-10-04 (Actual); Status verified 2017-10

CONDITIONS: Depression; Bipolar Disorder; Mood Disorders; Insulin Resistance; Depressive Disorder, Major; Depressive Disorder
MeSH Terms: conditions — Depression; Bipolar Disorder; Mood Disorders; Insulin Resistance; Depressive Disorder, Major; Depressive Disorder

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Optional buffy coat sample

SUMMARY:
The purpose of this study is to study the relationship between insulin and glucose action and neuropsychological functioning (memory, attention, general thinking abilities) in persons with depression.

ELIGIBILITY:
Inclusion Criteria:1)Willingness to sign the Human Subject Protection Consent Form prior to enrollment into the study.

2)Men and women ages 20 to 65 years of age. 3)Diagnosis of unipolar, non-psychotic, non-melancholic major depressive disorder (MDD) or depressive episode of bipolar disorder (Bipolar I, II or NOS), based on a Structured Clinical Interview for DSM-IV Axis I disorders (SCID) and confirmed by a psychiatrist.

4) Depression severity as defined by score of <17 on the 21-item Hamilton Rating Scale for Depression and no psychiatric admission within 6 months from study entry and no suicide attempt within the last 12 months.

5)Adequate visual and auditory acuity to allow neuropsychological testing. 6)Stable regime of psychiatric medications for 1 month prior to insulin test. Exclusion Criteria:1)Diagnosis of possible or probable cognitive impairment.

2)For women only: pregnancy, breastfeeding. 3)Personal history of Type I or Type II diabetes. 4) Unstable cardiovascular disease or other major medical condition, or history of myocardial infarction within the previous year.

5)Significant cerebrovascular disease, as evidenced by neurological examination, uncontrolled hypertension (systolic blood pressure > 170 or diastolic blood pressures > 100).

6) Current drug or alcohol abuse. 7)History of neurological disorder, e.g. multiple sclerosis, stroke etc. 8)Use of any drug that may significantly affect psychometric testing, or the insulin testing

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Men and women ages 20 to 65 years of age of any ethnic background, with a diagnosis of depression, and whose depressive symptoms are currently in remission
Sampling Method: Non-Probability Sample
Enrollment: 57 (Actual)
Dates: Start 2009-07; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
To quantify insulin-mediated glucose uptake as assessed by the SSPG concentration in patients with depression and compare the values to those previously obtained in a healthy age-matched control population | Within 3 hours of initial infusion

SECONDARY OUTCOMES:
To examine the association between insulin resistance and cognitive performance and clinical course of depression in patients with depression | 1 wk

CONTACTS AND LOCATIONS:
Overall Officials: Dr Natalie Rasgon, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

REFERENCES:
- [Derived] Wroolie TE, Kenna HA, Singh MK, Rasgon NL. Association between insulin resistance and cognition in patients with depressive disorders: exploratory analyses into age-specific effects. J Psychiatr Res. 2015 Jan;60:65-72. doi: 10.1016/j.jpsychires.2014.10.001. Epub 2014 Oct 14. PMID 25455511
- See also: Stanford Center for Neuroscience in Women's Health — http://womensneuroscience.stanford.edu/